CLINICAL TRIAL: NCT06238882
Title: A Phase III Study Comparing Concurrent Nitroglycerin With Radiation Therapy vs Radiation Therapy Alone in Patients With Non-small Cell Lung Cancer With EGFR Mutations and Brain Metastases.
Brief Title: Nitroglycerin Plus Radiotherapy Versus Conventional Radiotherapy in Patients With Lung Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Head of Thoracic Oncology Unit, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (023/013/ICI)(CEI/083/22)
Record Dates: First submitted 2024-01-22; First posted 2024-02-02 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer; Brain Metastases; EGFR Gene Mutation
Keywords: Radiation therapy; Nitroglycerin; Brain metastases; EGFR mutation; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will be given patches of nitroglycerin during treatment with radiation therapy (30 Gy in 10 fractions, i.e. 10 days of treatment).
  Interventions: Combination Product: Nitroglycerin
- Control (No Intervention): Patients will be given a conventional treatment with radiation therapy (30 Gy in 10 fractions, i.e. 10 days of treatment).

INTERVENTIONS:
Combination Product: Nitroglycerin — Patients in the intervention group will receive four 8mg-patches (36 mg final dose) of transdermal nitroglycerin with 10 mg release in 24 hours, for 24 hours with 12-hour rest intervals (to avoid receptor saturation) during treatment with radiation therapy (30 Gy in 10 fractions, or 10 days of treatment).
  Other Names: Minitran® Patch
  Arms: Intervention

SUMMARY:
The goal of this interventional phase III clinical trial is to evaluate objective intracranial response rate (iORR) after a treatment with total cranial radiation therapy plus concomitant transdermal nitroglycerin (NTG) addition or total cranial radiation therapy only in patients with stage IV non-small cell lung cancer with brain metastases and EGFR mutation. The main questions it aims to answer are:

Determine progression-free survival (PFS) to CNS and overall survival (OS). Evaluate and compare the quality of life (QoL) of patients during and after treatment.

Evaluate the cognitive function of patients before, during and after treatment. Evaluate treatment-associated toxicity to grade adverse treatment events Evaluation of HIF1α, VEGF and ROS1 in peripheral blood before and after nitroglycerin treatment.

All participants will have laboratory tests at the beginning and end of radiation therapy. Cranial MRI will be performed prior to treatment and 12 weeks after the end of treatment, then every 16 weeks until intracranial progression. Patients in the interventional group will be given 36 mg patches of transdermal nitroglycerin for 24 hours with a 12-hour rest interval during treatment with radiation therapy. The control group will only receive total cranial radiation therapy at the same doses and with the same schedule.

DETAILED DESCRIPTION:
The prognosis of patients with central nervous system (CNS) metastases is poor. About 50% of patients with CPCNP and EGFR mutation have tumor activity in the central nervous system during the first 2 years of diagnosis.

Treatment with total cranial radiation therapy (CRT) has shown to have a benefit in local response and patient survival. However, resistance factors such as intratumoral hypoxia decrease the response by CRT.

Thus, the use of nitric oxide generators, such as nitroglycerin, has been shown to avoid radio resistance. A previous study conducted at our Institute showed that the addition of transdermal nitroglycerin (NTG) CRT increases intracranial response evaluated by objective radiological response in patients with NSCLC and the subgroup in which a greater benefit was seen was in patients with mutations in the EGFR gene.

In this study we propose that the addition of transdermal nitroglycerin to patients with brain metastases and mutations in the EGFR gene receiving CRT will have an increase in intracranial objective response.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced non-small cell lung cancer (which includes de novo stage IIIB-IV, according to the 8th edition AJCC, or recurrent disease), documented by histology and/or cytology.
* Presence of brain metastases, candidates for treatment with holocranial radiation therapy.
* Documented EGFR sensitivity mutation.
* Disease measurable by criteria: The Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM).
* 18 years and up.
* Functional status, by ECOG scale 0-2
* Life expectancy at least 12 weeks.
* Not receive vasodilator treatment as calcium channel blockers.
* Electrocardiogram
* Neutrophil count 1.5 x 103/mm3, platelet count >100 x (103/mm3).
* Serum bilirubin should be 1.5 of the upper normal limit (ULN, upper normal limit).
* AST and/or ALT 2 ULN (or 5 x ULN in patients with liver metastases).
* Serum creatinine 1.5 (ULN), or creatinine clearance 60ml/min.
* Ability to comply with study and follow-up procedures.
* Informed written (signed) consent to participate in the study.
* Have tumor tissue (paraffin blocks from diagnostic biopsy) obtained before systemic treatment

Exclusion Criteria:

* Any unstable systemic disease (including active infection, grade 4 hypertension, unstable angina, congestive heart failure, ischemic heart disease, liver, kidney disease).
* Patients with a history of allergy to glyceryl tinistate
* Any other malignant pathology within the previous 5 years (except for cervical carcinoma in situ or basal-cell skin cancer, treated appropriately).
* Pregnant and/or breastfeeding women.
* Meningeal carcinomatosis corroborated by cytopathological study.

Disposal Criteria:

* Failure to follow protocol rules.
* Loss of patient follow-up.
* Patients who express their desire not to continue the study.
* Patients with unacceptable toxicity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
iORR | From date after radiation treatment until the first documented progression date, or last evaluable assessment in the absence of progression, or death from any cause, whichever comes first, to 12 weeks of follow up.
  Objective intracranial response rate (iORR) in patients with lung cancer and brain metastases treated with total cranial radiation therapy plus concomitant transdermal nitroglycerin addition versus patients treated with total cranial radiation therapy only.

SECONDARY OUTCOMES:
iPFS | From date of treatment initiation until date of disease progression or worsening until 12 weeks, and every 16 weeks of follow up until progression.
  Intracranial progression-free survival (iPFS) in patients with lung cancer and brain metastases treated with total cranial radiation therapy plus concomitant transdermal nitroglycerin addition versus patients treated with total cranial radiation therapy only.
OS | Duration of patient survival from the date of treatment initiation until until 12 weeks, and every 16 weeks of follow up
  Overall survival (OS) in patients with lung cancer and brain metastases treated with total cranial radiation therapy plus concomitant transdermal nitroglycerin addition versus patients treated with total cranial radiation therapy only.
QoL | A day before, within, and a day after the date of treatment initiation until date of disease progression or worsening or 12 weeks, and every 16 weeks of follow up.
  Quality of Life (QoL) measured by EORTC QLQ C30/LC13 in patients with lung cancer and brain metastases treated with total cranial radiation therapy plus concomitant transdermal nitroglycerin addition versus patients treated with total cranial radiation therapy only.
  The EORTC QLQ-C30 questionnaire consists of 30 questions with five functional scores (physical, role, cognitive, emotional and social); a global health status score three symptom scale score (fatigue, pain, nausea and vomiting); and six independent one-it.
  All scale and single-item scores can be linearly transformed to a score ranged from 0 to 100. A higher score of global health and functional subscriptions indicates better functioning.
Cognitive function | A day before, within, and a day after the date of treatment initiation until date of disease progression or worsening or 12 weeks, and every 16 weeks of follow up.
  Evaluate the cognitive function of patients with lung cancer and brain metastases treated with nitroglycerin vs radiation therapy alone before, during and after treatment using the Neuropsi Attention and Memory (NAM) instrument.
  NEUROPSI evaluates attention, memory, and learning functioning in Spanish speakers.
  Subtests are organized into summary scores that yield a General Attention and Memory Index Score, an Attention Index, Memory Index, and each of the subtests.
  Subtests evaluate Orientation, Attention and Concentration, Working Memory, Immediate Verbal Memory, Delayed Verbal Memory, Immediate Visual Memory, Delayed Verbal Memory, and Executive Functions.
  The Neuropsi Attention and Memory includes theoretical updates and new test scores indexes. It includes an adjustment of the norms of Total Attention and Executive Functions and Total Attention and Memory according to the modification of the tasks of digit detection and Stroop test.
Treatment-related Toxicity | Thee date of day 1, 7 and 10 of therapy and the date of 12 weeks after treatment.
  Treatment-related toxicity in patients with lung cancer and brain metastases treated with total cranial radiation therapy plus concomitant transdermal nitroglycerin addition versus patients treated with total cranial radiation therapy only using NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 to grading adverse events (AE).
  A grading (severity) scale is provided for each AE term. The CTCAE displays Grades 1 through 5:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental ADL*.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL**.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta, M.D., M.Sc., Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico